## Cover page

## **Statistical Analysis Plan**

## Official title of study:

Effect of Topical Lidocaine on Warm and Cold Sensation in Healthy Individuals - a Randomized Crossover Trial

NCT Number: 1-10-72-20-21

Document date: March 01, 2021

## Statistic TLH

Effect of Topical Lidocaine on Warm and Cold Sensation in Healthy Individuals

Endpoint Description of endpoint Statistic

Number PHS responders, original TSL, lidocaine compared to

Primary control McNemar

Secondary Number of TGI responders, lidocaine compared to control. McNemar

Strength of the TGI between TGI and non-TGI control stimuli

cold paired t-test/Wilcoxon

warm paired t-test/Wilcoxon

unpleasantness rating paired t-test/Wilcoxon

pain rating paired t-test/Wilcoxon

Number of PHS and TGI responses at baseline, i.e. without any

treatment McNemar

**Tertiary** 

QST active vs control

CDT paired t-test/Wilcoxon WDT paired t-test/Wilcoxon

CPT paired t-test/Wilcoxon HPT paired t-test/Wilcoxon

MDT paired t-test/Wilcoxon MPT paired t-test/Wilcoxon

Number of PHS responders using the TSL\_QST vs mTSL McNemar

nTSL

warm detection threshold when warming or cooling the skin

prior to test vs baseline paired t-test/Wilcoxon

cold detection threshold when warming or cooling the skin prior

to test vs baseline paired t-test/Wilcoxon

Number of PHS when warming or cooling the skin prior to test vs

baseline McNemar